CLINICAL TRIAL: NCT02090166
Title: Lung Cancer Detection and Staging by Extracellular Monitoring of Metabolic Activity Profiles of Peripheral Blood Mononuclear Cells (PBMC)
Brief Title: Lung Cancer Detection by Measuring Monocyte Activity
Acronym: EDLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-13-0105-CTIL
Record Dates: First submitted 2014-03-10; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lung cancer diagnosis (Other): 4 arms will be included in the study:
  The groups sample size is as follows:
  Group 1 - Healthy non smoker- 75 subjects Group 2 - Healthy smoker- 75 subjects Group 3 - Patients diagnosed as having COPD- 150 subjects Group 4 - Patients with diagnosis of lung cancer- 650 subjects
  A blood test will be taken from each patient.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — a blood test will be taken from each patient

SUMMARY:
Purpose: To evaluate the performance of Extracellular Monitoring of Metabolic Activity Profiles of Peripheral Blood Mononuclear Cells (PBMC) analysis method in identifying lung cancer.

The study population will include a total of 950 participants, patients with lung cancer before any treatment, and healthy and COPD patients as a control group.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the performance of Extracellular Monitoring of Metabolic Activity Profiles of Peripheral Blood Mononuclear Cells (PBMC) analysis method in identifying lung cancer.

The analysis method described in this protocol is a novel simple plausible immunological approach which is non-invasive, high throughput, real-time quantitative monitoring of metabolic activity (MA) profiles of fresh Peripheral Blood Mononuclear Cells (PBMC) in response to various reagents at different concentrations.

Study Design Prospective, three groups, open, comparative, controlled study. No. of Sites One Study Population Man and Women aged 18 - 90 years old. No. of Subjects A total of 950 completed, evaluated subjects will be enrolled in this study.

The groups sample size is as follows:

Group 1 - 75 subjects Group 2 - 75 subjects Group 3 - 150 subjects Group 4 - 650 subjects

Primary End Point 1. Positive and negative diagnosis (scored 0/1 dichotomously) in accordance with clinical data collected

Data Analysis and Statistics Multiple MA profiles including a huge number of MA rates values are obtained for each subject. In order to develop a dynamic clinical analysis that is updated with every new subject, and to extract patterns from this large data base, The research team designed computer programming using Data Mining tools, which combine methods from statistics and artificial intelligence with database management.

Blood test will be perform from each subject. The blood sample in eah subject will be compare to his status : healthy non smoker, healthy smoker, COPD or diagnosed with lung cancer.

ELIGIBILITY:
Inclusion Criteria

1. Subject signed the informed consent.
2. Subject is between 18 to 90 years old.
3. Lung cancer diagnosis before any treatment

Exclusion Criteria

1. Lung cancer patients
2. Subject has been previously treated for any type of malignant or benign tumor (for example: colon or uterus polyps removal).
3. Subject has active infection or inflammation determined clinically at screening.
4. Subject is currently treated with concomitant medication related directly or can affect the immune system.
5. Subject lactating or undergoing fertility treatment.
6. Subject has impaired judgment.
7. Known positive HIV, hepatitis B, or hepatitis C, autoimmune disease.
8. Known history of a significant medical disorder, which in the investigators' judgment contraindicates the patient's participation.
9. Known hypersensitivity and/or allergy
10. Drug or alcohol abuse (by history).
11. Subject is participating in any other clinical trial, drug or device study within 30 days prior sample collection
12. Relatives of the study investigators or employees of the study investigators are not allowed to participate in the study

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Positive and negative diagnosis (scored 0/1 dichotomously) of lung cancer | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Adir, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel